CLINICAL TRIAL: NCT00616044
Title: Continuous Spinal Anesthesia Versus Combined Spinal Epidural Block for Major Orthopedic Surgeries. Study Prospective and Randomized.
Brief Title: Continuous Spinal Anesthesia Versus Combined Spinal Epidural Block
Acronym: Spinocath
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sao Jose do Rio Preto Medical School (Other)
Responsible Party: Luiz Eduardo Imbelloni, MD. Director of Institute Regional Anesthesia, Hospital de Base, São José do Rio Preto, São Paulo, Brazil., Hospital de Base, São José do Rio Preto, São Paulo, Brazil.
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Imbelloni&Gouveia; Not applied
Record Dates: First submitted 2008-02-04; First posted 2008-02-15 (Estimated); Last update posted 2008-02-15 (Estimated); Status verified 2008-01

CONDITIONS: Hip Fractures; Knee Arthroplasty; Femur Fracture
Keywords: Spinal Anesthesia; Epidural Anesthesia; Orthopedic procedures
MeSH Terms: conditions — Hip Fractures; Femoral Fractures | interventions — Catheters

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- CSA (Experimental): For CSA, an 22-G catheter (Spinocath, B.Braun Melsungen, Germany) over a 27-G Quincke needle was used. After identification of the epidural space with a Crawford needle, the catheter with the spinal needle inside was advanced through the epidural space until the dural puncture was felt and CSF was seen in the catheter. The catheter was then fed over the needle into the intrathecal space. The spinal needle and the modified Tuohy needle were removed and a luer connector and a filter previously filled with the anesthetic solution were attached to the catheter.
  Interventions: Procedure: continuous spinal anesthesia; Procedure: Spinocath a catheter for continuous spinal anesthesia
- CSE (Experimental): CSE was performed with the "needle-through-needle" technique using a single interspace (Espocan, B.Braun Melsungen, Germany). The block consists of performing a spinal block via a 27-G spinal needle (Spinocan 125mm) introduced through an 18-G Tuohy needle (Perican 88mm) which was placed cranially directed in the epidural space. We did rotate the Tuohy needle between the spinal block and the insertion of the epidural catheter.
  Interventions: Procedure: Spinocath a catheter for continuous spinal anesthesia; Procedure: combined spinal epidural anesthesia

INTERVENTIONS:
Procedure: continuous spinal anesthesia — bupivacaina isobaric 0.5%, 5 mg
  Other Names: Major orthopedic surgeries
  Arms: CSA
Procedure: Spinocath a catheter for continuous spinal anesthesia — Continuous spinal anesthesia with low dose of bupivacaine isobaric Combined epidural spinal anesthesia with low dose of bupivacaine isobaric
  Other Names: Catheter for continuous spinal anesthesia; Catheter for combined spinal epidural anesthesia
Procedure: combined spinal epidural anesthesia — CSE was performed with the needle-through-needle technique using a single interspace (Espocan, B.Braun Melsungen, Germany
  Other Names: Catheter for continuous spinal anesthesia; Catheter for combined spinal epidural anesthesia
  Arms: CSE

SUMMARY:
In major orthopaedic surgery of the lower extremities both continuous spinal anesthesia (CSA) and combined spinal epidural anesthesia (CSE) are safe and reliable anaesthesia methods. Our results suggest that both continuous spinal anesthesia and combined spinal epidural anesthesia provide good surgical conditions with a low incidence of complications. The sensory block level and hemodynamic changes were lesser with CSA.

DETAILED DESCRIPTION:
240 patients scheduled for hip, knee arthroplasty or fracture of the femur were randomly assigned to receive either CSA or CSE. Blocks were performed in the lateral position at L3-L4 interspace. Puncture success, technical difficulties, paresthesia, highest level of sensory and motor block, need for complementary doses of local anesthetic, degree of technical difficulties, cardiocirculatory changes and post dural puncture headache were registered. At the end of the surgery, the catheter was removed and CSF leak was evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Fractures repair of femur, or arthroplasty of either knee or hip

Exclusion Criteria:

* Hypovolemia
* Preexisting neurologic disease
* Coagulation disorders and/or administration of thromboprophylaxis less than eight hours before the start of surgery
* Infection at the puncture site
* Agitation or delirium and the presence of a urinary bladder catheter.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2008-03; Primary Completion 2008-02 (Estimated); Study Completion 2009-01 (Estimated)

PRIMARY OUTCOMES:
Comparison between continuous spinal anesthesia versus combined spinal-epidural anesthesia in major orthopedic surgeries. | five years

CONTACTS AND LOCATIONS:
Overall Officials: Luiz E Imbelloni, MD, Principal Investigator — Sao Jose do Rio Preto Medical School
Locations (1):
- SaoJoseRPU, São José do Rio Preto, São Paulo, Brazil